CLINICAL TRIAL: NCT05817097
Title: Effect of Dipeptidyl-4 Inhibitors in Reducing Stroke Severity, From the Health Insurance Review and Assessment Service Database
Brief Title: Effect of Dipeptidyl-4 Inhibitors in Reducing Stroke Severity, From HIRA Database
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Seong-Joon Lee, Assistant professor, Ajou University School of Medicine
Other Study IDs: AJOUIRB-EX-2023-089
Record Dates: First submitted 2023-03-08; First posted 2023-04-18 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cerebral Infarction; Infarction, Brain; Dipeptidyl-Peptidase IV Inhibitors
Keywords: Dipeptidyl-Peptidase IV Inhibitors; Antidiabetic Drug
MeSH Terms: conditions — Cerebral Infarction; Brain Infarction | interventions — Dipeptidyl-Peptidase IV Inhibitors; 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- DPP4i: used DPP-4 inhibitors as anti-diabetic drugs before cerebral infarction(requiring thrombolysis or endovascular recanalization) Combination therpay is acceptable.
  Interventions: Drug: Dipeptidyl peptidase-4 inhibitor
- except DPP4i: patients that did not use DPP-4 inhibitors as anti-diabetic drugs before cerebral infarction(requiring thrombolysis or endovascular recanalization)

INTERVENTIONS:
Drug: Dipeptidyl peptidase-4 inhibitor — The definition of antidiabetic drug use is defined as a case in which an antidiabetic drug was prescribed for at least 2 months before stroke and the duration of treatment for stroke coincided with the prescribed duration of the drug.
  Other Names: A10BH07; EVOGLIPTIN; Suganon Tab
  Groups: DPP4i

SUMMARY:
The goal of this observational study is to compare severity and mortality rates of acute cerebral infarction(requiring thrombolysis or endovascular recanalization) depending on the type of oral antidiabetic drug taken before the onset of cerebral infarction.

Researchers will compare the group that used DPP-4 inhibitors as anti-diabetic drugs before cerebral infarction and the group that did not use them to see the effect of DPP-4 inhibitors in reducing severity of cerebral infarction.

DETAILED DESCRIPTION:
This is a retrospective study to see the effects of reducing the severity of cerebral infarction(requiring thrombolysis or endovascular recanalization) of DPP-4 inhibitors by comparing the survival rate after acute cerebral infarction hospitalization, discharge rate to home, and medical cost.

A. Severity of cerebral infarction and poor prognosis is mainly associated with hyperglycemia caused by diabetes, which increases the Infarction volume and hemorrhagic trasformation.

B. However, the effect of loergin blood glucose on reducing the Infarction volume and improving prognosis of cerebral infarction has not been proven.

C. Preclinical studies have demonstrated a anti-stroke effect that reduces the Infarction volume using certain anti-diabetic drugs.

D. Therefore, there is a possibility that certain anti-diabetic drugs may reduce the severity of cerebral infarction as a class effect in addition to the effect of blood sugar control.

E. This is particularly likely to exist in the DPP-4 inhibitor family identified through preclinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute cerebral infarction who underwent thrombolysis or endovascular recanalization in Korea between 2014 and 2021
* Those who have been previously diagnosed with diabetes and are taking oral anti-diabetic drugs
* Adult (over 19 years of age)

  * The definition of antidiabetic drug use is defined as a case in which an antidiabetic drug was prescribed for at least 2 months before stroke and the duration of treatment for stroke coincided with the prescribed duration of the drug.

Exclusion Criteria:

* Patients taking insulin to control diabetes

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study using the Health Insurance Review and Assessment Service (HIRA) database in Korea.
  In this database, patients with acute cerebral infarction who underwent thrombolysis(intravenous thrombolysis) or endovascular recanalization (intraarterial thrombectomy) between 2014 and 2021 is included.
Sampling Method: Probability Sample
Enrollment: 22119 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | Check the data one year after the onset of stroke.
  The survival rates of the DPP-4 inhibitor group and the non-use group are compared 1 year after the onset of severe stroke.
90-day survival rate | Check the data 90-day after the onset of stroke.
  The survival rates of the DPP-4 inhibitor group and the non-use group are compared 90-day after the onset of severe stroke.
re-hospitalization | 1 year after discharge the stroke treatment.
  The re-hospitalization rates of the DPP-4 inhibitor group and the non-use group are compared after the onset of severe stroke.
frequency of cerebral hemorrhage | Hospitalization period and 1 year after discharge the stroke treatment.
  The frequency of cerebral hemorrhage rates of the DPP-4 inhibitor group and the non-use group are compared after the onset of severe stroke.
Rate of Intensive care unit treatment | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The Intensive care unit treatment rate of the DPP-4 inhibitor group and the non-use group are compared.
Duration of Intensive care unit | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The duration of Intensive care unit of the DPP-4 inhibitor group and the non-use group are compared.
Rate of Stroke care unit treatment | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The Stroke care unit treatment rate of the DPP-4 inhibitor group and the non-use group are compared.
Duration of Stroke care unit | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The duration of Stroke care unit of the DPP-4 inhibitor group and the non-use group are compared.
tracheal intubation period | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The tracheal intubation period of the DPP-4 inhibitor group and the non-use group are compared.
total hospitalization days | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The total hospitalization days of the DPP-4 inhibitor group and the non-use group are compared.
medical expenses incurred at the time of hospitalization | Hospitalization period is expected to be up to three months. It is not possible to accurately estimate the period of hospitalization due to severe stroke.
  The medical expenses incurred at the time of hospitalization of the DPP-4 inhibitor group and the non-use group are compared.

SECONDARY OUTCOMES:
Home discharge rate | At the end of discharge from stroke treatment.
  The Home discharge rate of the DPP-4 inhibitor group and the non-use group are compared.
medical expenses after discharge from hospital | 1 year after discharge the stroke treatment.
  The medical expenses after discharge from hospital of the DPP-4 inhibitor group and the non-use group are compared.

CONTACTS AND LOCATIONS:
Overall Officials: DukYong Yoon, MD., PhD., Principal Investigator — Department of Biomedical Systems Informatics,Yonsei University College of Medicine,Yongin,SouthKorea; Seong-Joon Lee, MD., PhD., Principal Investigator — Department of Neurology, Ajou University School of Medicine, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No
Ajou University Hospital's IRB(Institutional Review Board) sends IRB approval documents to HIRA and conducts research with anonymized data after request.
  Data collected during the research process will be stored for 3 years and then properly disposed of in accordance with relevant laws.

REFERENCES:
- [Result] Sinha B, Ghosal S. Meta-analyses of the effects of DPP-4 inhibitors, SGLT2 inhibitors and GLP1 receptor analogues on cardiovascular death, myocardial infarction, stroke and hospitalization for heart failure. Diabetes Res Clin Pract. 2019 Apr;150:8-16. doi: 10.1016/j.diabres.2019.02.014. Epub 2019 Feb 20. PMID 30794833
- [Result] Darsalia V, Ortsater H, Olverling A, Darlof E, Wolbert P, Nystrom T, Klein T, Sjoholm A, Patrone C. The DPP-4 inhibitor linagliptin counteracts stroke in the normal and diabetic mouse brain: a comparison with glimepiride. Diabetes. 2013 Apr;62(4):1289-96. doi: 10.2337/db12-0988. Epub 2012 Dec 3. PMID 23209191
- [Result] Lee SJ, Yoon BS, Hong JM, Joe EH, Lee JS. Effects of co-administration of metformin and evogliptin on cerebral infarct volume in the diabetic rat. Exp Neurol. 2022 Feb;348:113922. doi: 10.1016/j.expneurol.2021.113922. Epub 2021 Nov 12. PMID 34780772
- [Result] Johnston KC, Bruno A, Pauls Q, Hall CE, Barrett KM, Barsan W, Fansler A, Van de Bruinhorst K, Janis S, Durkalski-Mauldin VL; Neurological Emergencies Treatment Trials Network and the SHINE Trial Investigators. Intensive vs Standard Treatment of Hyperglycemia and Functional Outcome in Patients With Acute Ischemic Stroke: The SHINE Randomized Clinical Trial. JAMA. 2019 Jul 23;322(4):326-335. doi: 10.1001/jama.2019.9346. PMID 31334795
- [Result] Kim JY, Kang K, Kang J, Koo J, Kim DH, Kim BJ, Kim WJ, Kim EG, Kim JG, Kim JM, Kim JT, Kim C, Nah HW, Park KY, Park MS, Park JM, Park JH, Park TH, Park HK, Seo WK, Seo JH, Song TJ, Ahn SH, Oh MS, Oh HG, Yu S, Lee KJ, Lee KB, Lee K, Lee SH, Lee SJ, Jang MU, Chung JW, Cho YJ, Choi KH, Choi JC, Hong KS, Hwang YH, Kim SE, Lee JS, Choi J, Kim MS, Kim YJ, Seok J, Jang S, Han S, Han HW, Hong JH, Yun H, Lee J, Bae HJ. Executive Summary of Stroke Statistics in Korea 2018: A Report from the Epidemiology Research Council of the Korean Stroke Society. J Stroke. 2019 Jan;21(1):42-59. doi: 10.5853/jos.2018.03125. Epub 2018 Dec 18. PMID 30558400
- [Result] Park SH, Jeong HE, Oh IS, Hong SM, Yu SH, Lee CB, Shin JY. Cardiovascular safety of evogliptin in patients with type 2 diabetes: A nationwide cohort study. Diabetes Obes Metab. 2021 Jun;23(6):1232-1241. doi: 10.1111/dom.14330. Epub 2021 Feb 10. PMID 33502058
- [Result] Shim DH, Kim Y, Roh J, Kang J, Park KP, Cha JK, Baik SK, Kim Y. Hospital Volume Threshold Associated with Higher Survival after Endovascular Recanalization Therapy for Acute Ischemic Stroke. J Stroke. 2020 Jan;22(1):141-149. doi: 10.5853/jos.2019.00955. Epub 2020 Jan 31. PMID 32027799